CLINICAL TRIAL: NCT02902003
Title: Testing the Effectiveness of Offering Relationship Skills Education Services With a Robust Economic Security Component to Low-income Couples Raising Children.
Brief Title: Testing Relationship Skills Education Services With a Robust Economic Security Component
Acronym: TPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPR-500098-TPC
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Family Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Not eligible for program services
- Empowering Families (Active Comparator): These couples will be eligible to participate in the "Empowering Families" program.
  Interventions: Behavioral: Empowering Families

INTERVENTIONS:
Behavioral: Empowering Families — A program that integrates the healthy relationship curriculum, Family Wellness, into a comprehensive set of services that includes case management, employment services, and financial coaching. The program will have four core components: (1) 20 hours of core workshop sessions using the Family Wellness curriculum; (2) case management; (3) employment services; and (4) financial coaching. The core component of Empowering Families will be a 20-hour group workshop, organized into eight two-and-a-half-hour weekly sessions (Table 1). The main content of these sessions will be based on the Family Wellness relationship education curriculum which will be covered in six sessions. These six sessions will be led by two trained facilitators employed by The Parenting Center. The core workshops will be supplemented with two additional sessions on financial planning and employment topics that will designed to be useful to all participants, regardless of their level of financial and employment needs.
  Arms: Empowering Families

SUMMARY:
The Parenting Center (TPC) offers the Empowering Families program, which integrates a relationship education curriculum (Family Wellness) into a comprehensive set of services that includes case management, employment services, and financial coaching. The evaluation will test the effectiveness of offering relationship skills education services with a robust economic security component to low-income couples raising children.

DETAILED DESCRIPTION:
The evaluation of Empowering Families will test the effectiveness of offering relationship skills education services with a robust economic security component to low-income couples raising children. The program is built on Family Wellness, a relationship education curriculum that has not yet been rigorously studied. The Parenting Center (TPC) has integrated Family Wellness into a comprehensive set of services that includes case management, employment services, and financial coaching. The evaluation will test the effect of this full package of services on couples' relationship and employment outcomes. The evaluation will also examine effects on outcomes related to child well-being, such as co-parenting and father involvement.

The Empowering Families evaluation will be conducted with low-income couples raising children. To be eligible for program services, both members of the couple must: (1) be age 18 or older, (2) report that they are in a committed relationship with their partner; (3) speak a language in which programming is being offered; (4) be interested in participating in a program that offers both relationship skills and economic stability services; (5) be available to participate in programming for the next six months; (6) pass a domestic violence screen; and (7) not have an open case with child protective services. In addition, at least one member of the couple must have a biological or adopted child who is under age 18 and lives with them at least half time. The Parenting Center will aim to recruit couples who are economically disadvantaged and likely to want both relationship skills and employment services.

The evaluation plan for the Empowering Families program calls for the enrollment and random assignment of 1,000 couples over the course of two years. This target requires The Parenting Center to recruit approximately 42 couples for the study each month. Half of these couples will be randomly assigned to the Empowering Families program; the other half will be assigned to a control group that is not eligible for program services.To document the outcomes of study participants, survey data will be collected at two time points: (1) a baseline survey administered at study enrollment and (2) a follow-up survey conducted about a year later. The investigators will also conduct a process study to document how Empowering Families was implemented.

ELIGIBILITY:
Inclusion Criteria: (Necessary for eligibility)

1. age 18 or older
2. report that they are in a committed relationship with their partner
3. speak a language in which programming is being offered
4. be interested in participating in a program that offers both relationship skills and economic stability services
5. be available to participate in programming for the next six months;
6. pass a domestic violence screen
7. not have an open case with child protective services.
8. at least one member of the couple must have a biological or adopted child who is under age 18 and lives with them at least half time.

Exclusion Criteria:

* Ineligible if do not meet any of the above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1758 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Employed or taking steps to find a job | 1 year after random assignment
  a binary variable equal to 1 if a respondent was ever employed at any time during the first year after study enrollment or indicates that in the past year he/she has done any of the following:
  * Created or updated a resume
  * Looked for a job
  * Submitted a job application
  * Gone on a job interview
Monthly earnings | 1 year after random assignment
  This continuous variable uses survey data and is based on average monthly earnings from all jobs in the first year following study enrollment. It will be analyzed separately for men and women.
Family economic hardship scale | 1 year after random assignment
  This scale represents how many of six economic hardships the family experienced in the past year.
Quality of co-parenting relationship | 1 year after random assignment
  This 10-item scale (α = 0.94) is the average level of agreement-from "strongly disagree" (= 1) to "strongly agree" (= 4)-with statements about the respondent's partner, constructed by averaging across partners' responses.
Couple married to each other | 1 year after random assignment
  This is a binary variable equal to 1 if both partners report that they are married to each other
Couple married or romantically involved | 1 year after random assignment
  This is a binary variable equal to 1 if both partners report that they are married to each other or in a romantic relationship with each other
Support and affection | 1 year after random assignment
  This 12-item scale is the average level of agreement-from "strongly disagree" (= 1) to "strongly agree" (= 4)-with statements about the respondent's partner, constructed by averaging across partners' responses
Avoidance of destructive conflict behaviors | 1 year after random assignment
  This eight-item scale (α = 0.92) is the average frequency-from "never" (= 1) to "often" (= 4)-that a respondent reports experiencing destructive conflict behaviors with his or her partner, constructed by averaging across partners' responses
Constructive conflict behaviors | 1 year after random assignment
  This seven-item scale (α = 0.87) is the average frequency-from "never" (= 1) to "often" (= 4)-that a respondent reports experiencing constructive conflict behaviors with his or her partner, constructed by averaging across partners' responses
Relationship commitment | 1 year after random assignment
  This continuous variable ranges from 0 to 10, with higher values indicating that both partners are more committed to their romantic relationship. The measure is the average across the two partners' responses.
Relationship happiness | 1 year after random assignment
  This continuous variable ranges from 0 to 10, with higher values indicating that both partners report greater happiness with their romantic relationship. The measure is the average across the two partners' responses.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wood, PhD, Study Director — Mathematica Policy Research
Locations (1):
- The Parenting Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No